CLINICAL TRIAL: NCT01463748
Title: Effects of Graptopetalum Paraguayense E. Walther on the Oxidative Stress, Antioxidant Enzyme Activity and Inflammation in Subjects With Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chun-Yu Yeh, Assistant Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CS11074
Record Dates: First submitted 2011-10-31; First posted 2011-11-02 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): starch
  Interventions: Other: Placebo
- Graptopetalum paraguayense E. Walther (Experimental): Graptopetalum paraguayense E. Walther
  Interventions: Other: Graptopetalum paraguayense E. Walther

INTERVENTIONS:
Other: Graptopetalum paraguayense E. Walther — Graptopetalum paraguayense E. Walther
  Arms: Graptopetalum paraguayense E. Walther
Other: Placebo — starch
  Other Names: starch
  Arms: Placebo

SUMMARY:
Metabolic syndrome (MS) is a significant risk factor of cardiovascular disease. The purposes of this study are going to investigate the effects of Graptopetalum paraguayense E. Walther on the oxidative stress, antioxidant enzyme activity and inflammation in subjects with metabolic syndromerelation. The investigators will recruit MS patients(n=50)and the inclusion criteria of MS are according to the Bureau of Health Promotion, Department of Health in Taiwan (2007). The MS subjects are randomly assigned to placebo(n=25) and Graptopetalum paraguayense E. Walther supplements(n=25)groups. Hopefully, the results of this study could provide the information of Graptopetalum paraguayense E. Walther supplements to what has been know in MS subjects.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of MS in adult are according to the Bureau of Health Promotion, Department of Health in Taiwan (2007), if subjects had 3 of the following 5 characteristics: (1) abdominal obesity (waist circumference >= 90 cm in men and >= 80 cm in women), (2) impaired fasting glucose ( >= 5.6 mmol/L), (3) hypertriglyceridemia ( >= 1.7 mmol/L), (4) low HDL-C (< 1.0 mmol/L in men and < 1.3 mmol/L in women), and (5) increased blood pressure (SBP >= 130 mmHg and DBP >= 85 mmHg). Subjects using antidiabetic or antihypertensive or lipid-lowering medications were considered to have elevated fasting blood glucose or elevated blood pressures or dyslipidemia, respectively.

Exclusion Criteria:

* Subjects with liver, renal diseases, undergoing statin therapy, pregnancy women, and taking antioxidant vitamins supplements were excluded.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Antioxidant and inflammation | 12 weeks
  The study are going to measure the concentrations of lipid peroxidation markers (TBARS and ox-LDL) and antioxidant enzymes activities (catalase, glutathione peroxidase, and superoxide dismutase), and the level of inflammatory markers (hs-CRP, TNF-alfa, IL-1, IL-6 and adiponectin) in all subjects of this study.

SECONDARY OUTCOMES:
Blood biochemical values | 12 weeks
  Fasting glucose, blood pressure, and blood lipid profiles(total cholesterol, triglyceride, low density lipoprotein and high density lipoprotein).

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

REFERENCES:
- [Derived] Yen CH, Chen SJ, Liu JT, Tseng YF, Lin PT. Effects of water extracts of Graptopetalum paraguayense on blood pressure, fasting glucose, and lipid profiles of subjects with metabolic syndrome. Biomed Res Int. 2013;2013:809234. doi: 10.1155/2013/809234. Epub 2013 Nov 25. PMID 24371832